CLINICAL TRIAL: NCT03419221
Title: Impact of 18 FDG PET/CT on the Management of Patients With Staphylococcus Aureus Bloodstream Infection. An Open-comparative Randomized Trial
Brief Title: Impact of 18 FDG PET/CT on the Management of Patients With Staphylococcus Aureus Bloodstream Infection
Acronym: TEPSTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UF 9788
Record Dates: First submitted 2017-11-08; First posted 2018-02-01 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Staphylococcus Aureus
Keywords: Staphylococcus aureus; bloodstream infection; deep foci of infection; 18 FDG PET/CT; antibiotics
MeSH Terms: conditions — Staphylococcal Infections; Sepsis | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: Patients with PET/CT performs at day 14 after the drawing (Active Comparator): Arm A: Patients with PET/CT performs at day 14 after the drawing of the first blood culture
  Interventions: Procedure: PET/CT Positron emission tomography (PET) using small radiotracers, a special camera and a computer to evaluate organ and tissue functions
- B : Patients' routine care with performance of explorations (Placebo Comparator): Arm B : Patients' routine care with performance of explorations based on anamnesis and clinical symptoms
  Interventions: Other: Patients' routine care with performance of explorations based on anamnesis and clinical symptoms

INTERVENTIONS:
Procedure: PET/CT Positron emission tomography (PET) using small radiotracers, a special camera and a computer to evaluate organ and tissue functions — Open-label randomized controlled superiority trial in patients with SAB without infective endocarditis at the time of inclusion comparing whole-body PET/CT in arm A and routine care with performance of imaging studies according to anamnesis and clinical symptoms in arm B. To demonstrate that PET/CT is associated with a 20% higher frequency of detection of DFI during SAB, the inclusion of 145 patients in each arm is required.
  Randomization will be stratified on centre and SAB setting of acquisition (healthcare vs community).
  Arms: A: Patients with PET/CT performs at day 14 after the drawing
Other: Patients' routine care with performance of explorations based on anamnesis and clinical symptoms — Patients' routine care with performance of explorations based on anamnesis and clinical symptoms
  Arms: B : Patients' routine care with performance of explorations

SUMMARY:
S. aureus bloodstream infection (SAB) is a severe disease associated with a 30% case-fatality rate at 12 weeks. Severity of this disease is related to the high prevalence of staphylococcal Deep Foci of Infection (SA-DFI), which require prolonged duration of antimicrobial therapy and specific treatment. Timely diagnosis and management of SA-DFI is associated with an improvement of prognosis during SAB. 18 FDG PET/CT (PET/CT) is a useful tool in the diagnosis of infectious foci during bacterial infections.

An ecological study performed in the Netherlands has shown that use of PET/CT in patients with Gram positive cocci bloodstream infection was associated with an increase of detection of DFI and a decrease of recurrences and mortality compared to historical controls.

The investigators hypothesize that SAB poor prognosis is in part related to the lack of diagnosis of all infectious foci and consequently to a suboptimal treatment.

DETAILED DESCRIPTION:
Subjects will be recruited in medical wards of the 10 participating hospitals. Each included patient will be managed according to clinical expertise of investigators who all are experts in the field of infectious diseases. Consensual guidelines for antimicrobial therapy of patients enrolled in the study will be written before the enrolment of the first patient by the steering committee composed of all co-investigators These guidelines will specify the nature of empiric therapy as well as adapted antibiotic therapy for each specific DFI for methicillin-sensitive as well as for methicillin resistant S. aureus.

Experimental group: arm A All patients enrolled in arm A will have a PET/CT after enrolment and not later than day 14 after the drawing of first positive blood culture.

Control group: arm B Patients enrolled in arm B will not have PET/CT before day 14. Other imaging studies will be guided by anamnesis and clinical symptoms and performed according to guidelines written consensually before the enrolment of the first patient by the steering committee

ELIGIBILITY:
Inclusion Criteria:

* - Aged over 18 years
* Signed informed consent form
* Subjects must be able to attend all scheduled visits and to comply with all trial procedures
* Subjects must be covered by public health insurance
* Hospitalized in one of the 10 participating centres
* At least one peripheral blood culture isolating S. aureus
* Absence of diagnosis of IE according to at least a transthoracic cardiac echography; cardiac echography will be performed via transesophageal procedure if the VIRSTA score is 3 or higher (see Appendix) or if transthoracic echography is not normal.

Exclusion Criteria:

* - Any reason that may compromise compliance with the visit plan
* Planned longer stay outside the region that prevents compliance with the visit plan
* Deprived of liberty subjects (by judicial or administrative decision)
* Adult under guardianshipCatheter-related SAB with resolution of symptoms of infection within 24 hours of ablation of catheter
* Pregnancy or lactation
* Isolation of S. aureus only in blood cultures drawn from a catheter or another implanted device
* Catheter-related SAB with resolution of symptoms of infection within 24 hours of ablation of catheter
* Uncontrolled septic shock and other instability contra-indicating the performance of PET/CT
* Previous performance of PET/CT for the present episode of SAB
* Indication to PET/CT for another reason (eg. neoplasm, infection of vascular graft…)
* Contra-indication to PET/CT
* Contraindication to Fluorodeoxyglucose : hypersensitivity to the active substance or to any of the excipients
* Participation to another study unless specific authorization of the steering committee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Presence of at least one DFI following the drawing of the first blood positive culture. | day 14
  SA-DFI will be defined as the presence of at least one of the following criteria adapted form the criteria proposed by EMA for evaluation of antibiotics (EMA):
  * Deep collection without any other explanation than S. aureus infection
  * Osteomyelitis or arthritis without any other explanation than S. aureus infection; in case of presence of material (osteosynthesis or prosthetic joint) the presence of clinical symptoms or bacteriological confirmation will be required because the specificity of imaging including PET/CT is low
  * Isolation of S. aureus in a sterile site other than blood, urine or catheter (eg: pleura, cerebrospinal fluid, bone, synovial fluid, muscle…)

SECONDARY OUTCOMES:
PET/CT Evaluation :Frequency of SA-DFI | day 14
  Frequency of SA-DFI according to the investigator
PET/CT Evaluation :Time to detection | day 14
  Time to detection of DFI
Duration of Antibiotic treatment | 3 months
  Duration of antibiotic treatment
Duration of Antibiotic treatment | 6 months
  Duration of antibiotic treatment
frequency of Diagnostic procedures | 3 months
  frequency of procedures performed to treat SA-DFIs
frequency of Diagnostic procedures | 6 months
  frequency of procedures performed to treat SA-DFIs
Recurrences of S. aureus infection | 3 months
  Frequency of recurrences
Recurrences of S. aureus infection | 6 months
  Frequency of recurrences
Survival | 3 months
  Survival
Survival | 6 months
  Survival
Evaluation of the cost-effectiveness of strategies | 3 months
  Cost-effectiveness of strategies
Evaluation of the cost-effectiveness of strategies | 6 months
  Cost-effectiveness of strategies
Diagnostic procedures :Detection of endocardial hyperfixation | 3 months
  Detection of endocardial hyperfixation at PET/CT in arm A
Diagnostic procedures :Detection of endocardial hyperfixation | 6 months
  Detection of endocardial hyperfixation at PET/CT in arm A

CONTACTS AND LOCATIONS:
Overall Officials: Vincent LE MOING, Professor, Principal Investigator — Infectious Diseases department of CHU-Montpellier
Locations (1):
- Chu Gui de Chauliac, Montpellier, France